CLINICAL TRIAL: NCT05958251
Title: Umbilical Cord Stump Medication with a Topical Dermo Protective Powder Compared to Dry Care in Healthy Full-term and Near-term Newborns: a Two Centres Prospective Cohort Study
Brief Title: The Use of Arnica Montana in the Cicatrization of the Umbilical Cord
Status: Completed | Type: Observational
Sponsor: Ospedale Buon Consiglio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Giuseppe De Bernardo, Head of Department of Woman and Child, Ospedale Buon Consiglio Fatebenefratelli
Other Study IDs: 496/CE Lazio 1
Record Dates: First submitted 2023-07-04; First posted 2023-07-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-07

CONDITIONS: Umbilical Cord Issue
Keywords: newborn; umbilical cord care; arnica; complications; infections
MeSH Terms: conditions — Infections | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cicaben: Umbilical cord stump of the newborns was medicated by Cicaben ® (Orsana S.r.l.), a natural topical dermo-protective powder
  Interventions: Other: Cicaben
- Standard dry care: Umbilical cord stump of the newborns was medicated by standard dry care
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Other: Cicaben — Cicaben® powder is an association of special active ingredients for topical dermatological use with a healing, soothing and protective action (zinc oxide, magnesium oxide, corn starch, arnica montana extract, allantoin and undecylenic acid, arginine, glycine and proline, niacinamide).
  Groups: Cicaben
Other: Standard Care (in control arm) — Standard care
  Groups: Standard dry care

SUMMARY:
Neonatal infections are still one of the leading causes of mortality among newborns worldwide. For example, omphalitis is particularly common and can lead to the development of neonatal sepsis. This pathology more frequently affects developing countries, where hygienic conditions are often precarious, but the incidence of this disease should not be underestimated even in developed countries. Therefore, it is essential to properly care for the umbilical stump during the first days of life to prevent infections, both in the hospital and at home.

The complications related to poor hygiene of the umbilical stump can be more or less serious. Mild complications include wet stumps, purulent secretions, granulomas, or periumbilical erythema. The most serious complications involve infections of the umbilical cord stump which can manifest locally or systemically, causing respectively omphalitis or neonatal sepsis. Despite the numerous benefits that derive from proper umbilical cord care, the most suitable approach remains controversial and several modalities of care have been described.

The World Health Organization suggests two techniques depending on the neonatal mortality rate. In developed countries the use of dry cord care is recommended while in countries with a high neonatal mortality rate (>30 deaths/1000 live births) the topical application of antiseptics, such as chlorhexidine, is recommended. Recent studies have focused on the possible advantages of using natural products of plant origin, whose natural anti-inflammatory and dermal protective action is known. Among them, the anti-inflammatory, antibacterial and immunomodulatory properties of arnica montana have been studied and it has been shown that the use of a powder containing this plant extract reduces parental stress and drop time of the umbilical cord stump. However, there is little evidence demonstrating the lower rate of mild to moderate complications resulting from umbilical cord stump care with this product.

DETAILED DESCRIPTION:
Neonatal infections are still an important cause of neonatal deaths, worldwide infections are estimated as the cause 4% to 56% of all neonatal deaths. Among the possible points of entry for invasive bacteria in neonates, omphalitis represents an important risk factor for neonatal sepsis and death. Even if the risk of omphalitis may be greater in countries with limited resources and poor hygienic conditions, also in developed countries, where the incidence is considered rare, it must not be ignored (0.7%). Consequently, proper umbilical cord stump care during the first days of life (both in hospital and at home) shouldn't be overlooked to prevent possible complications. The complications of poor hygiene of the umbilical cord stump can be serious. Mild complications include wet cord stumps, purulent discharge, granulomas, or periumbilical erythema. Severe complications include cord stump infections, which may be localized as omphalitis or, after entry in the blood circulation, systemic (neonatal sepsis). Despite the known benefits of its correct execution, the care of umbilical cord stump remains controversial, and many different approaches are described. The World Health Organisation suggests two techniques depending on neonatal mortality rate. In developed countries it is recommended the use of dry cord stump care while in countries with high neonatal mortality rate (>30 deaths/1000 live births) it is recommended topical antiseptics application (such as chlorhexidine). Dry care consists in cleansing the cord stump with a neutral soap at birth and then keeping the cord stump dry, avoiding the immersion in water. In some centres it is recommended to apply a clean and dry gauze around the cord stump or to keep the cord stump outside the diaper. Dry care is an easy and economic technique, but parents must be accurately instructed to detect precociously possible signs of infection. Topical antiseptics application is recommended in countries where hygienic conditions are poor and neonatal mortality rate is higher. However, this practice is often widely adopted also in developed countries, where from one side no significant advantages are described and on the other side It may increase risk of sensibilization to contact dermatitis and burning. A Cochrane review published in 2013 found that the use of medications such as chlorhexidine may increase the cord stump separation time, but there is no evidence that it increases risk of mortality or infection. In developing countries many other methods are used, some of them described in literature: in Africa some mothers apply cow dung and/or oil on the umbilical cord stump in Nigeria some women apply mentholated balm or toothpaste on the umbilical cord stump; mustard oil and turmeric are used in other regions. These techniques are mostly based on cultural traditions and derive both from a lack of healthcare in the perinatal period and from ignorance of the population regarding the correct standards of care. These methods are not recommended for a demonstrated increased risk of infection by C. tetani.The best management of umbilical cord stump care is still unknown. Recent studies investigated the use, in addition to dry care, of plant-derived topical products, which are known to have natural anti-inflammatory and dermo protective qualities. However, there is currently little evidence about their safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

Gestational age > 35 weeks and hospitalization in Standard Neonatal Care.

Exclusion Criteria:

* They were excluded newborns admitted in Neonatal Intensive Care Unit.

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: They were enrolled infants born in two centers: V. Buzzi Children's Hospital and Fatebenefratelli Hospital, ASST-FBF Sacco, Milan, Italy and Ospedale Buon Consiglio Fatebenefratelli, Naples, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Cicaben ® medication on the detachment of the umbilical cord stump | 48 hours after discharge
  Umbilical cord stump detachment will be evaluated by medical examination
Evaluation of the Cicaben ® medication on the presence of dry or wet umbilical cord stump | 48 hours after discharge
  The presence of dry or wet umbilical cord stump will be evaluated by medical examination
Evaluation of umbilical cord stump medication with Cicaben ® on mild complications | 48 hours after discharge
  Mild complications will be evaluated by medical examination
Evaluation of umbilical cord stump medication with Cicaben ® on periumbilical erythema | 48 hours after discharge
  Periumbilical erythema will be evaluated by medical examination
Evaluation of umbilical cord stump medication with Cicaben ® on purulent secretions | 48 hours after discharge
  Purulent secretions will be evaluated by medical examination
Evaluation of umbilical cord stump medication with Cicaben ® on granuloma | 48 hours after discharge
  Granuloma will be evaluated by medical examination
Evaluation of umbilical cord stump medication with Cicaben ® on the use of H2O2 and topical treatment with silver nitrate | 48 hours after discharge
  The use of H2O2 and topical treatment with silver nitrate will be evaluated by medical examination

SECONDARY OUTCOMES:
Evaluation of the Cicaben ® medication on the detachment of the umbilical cord stump | 1 week after discharge
  Umbilical cord stump detachment will be evaluated by medical examination
Evaluation of the Cicaben ® medication on the presence of dry or wet umbilical cord stump | 1 week after discharge
  The presence of dry or wet umbilical cord stump will be evaluated by medical examination
Evaluation of umbilical cord stump medication with Cicaben ® on mild complications | 1 week after discharge
  Mild complications will be evaluated by medical examination
Evaluation of umbilical cord stump medication with Cicaben ® on periumbilical erythema | 1 week after discharge
  Periumbilical erythema will be evaluated by medical examination
Evaluation of umbilical cord stump medication with Cicaben ® on purulent secretions | 1 week after discharge
  Purulent secretions will be evaluated by medical examination
Evaluation of umbilical cord stump medication with Cicaben ® on granuloma | 1 week after discharge
  Granuloma will be evaluated by medical examination
Evaluation of umbilical cord stump medication with Cicaben ® on the use of H2O2 and topical treatment with silver nitrate | 1 week after discharge
  The use of H2O2 and topical treatment with silver nitrate will be evaluated by medical examination

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe De Bernardo, MD, Principal Investigator — Ospedale Buon Consiglio Fatebenefratelli
Locations (2):
- Italy (2):
  - Vittore Buzzi Children's Hospital, ASST-FBF-Sacco, Milan, Milan
  - Ospedale Buon Consiglio Fatebenefratelli, Naples, Naples

IPD SHARING:
Plan to Share IPD: No